CLINICAL TRIAL: NCT03991741
Title: Phase I Trial of Lymphodepletion Followed by Adoptive Cell Transfer of Autologous Tumor Infiltrating Lymphocytes and High-Dose Interleukin 2 in Select Solid Tumors
Brief Title: Adoptive Cell Transfer of Autologous Tumor Infiltrating Lymphocytes and High-Dose Interleukin 2 in Select Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed because of feasibility and safety issues, didn't reach our end point
Sponsor: Gregory Daniels (Other)
Collaborators: Immunotherapy Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Gregory Daniels, Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160710
Record Dates: First submitted 2019-04-10; First posted 2019-06-19 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Melanoma; Locally Advanced Refractory/Recurrent Melanoma; Metastatic Head and Neck Cancer; Locally Advanced Refractory/Recurrent Head and Neck Cancer
Keywords: melanoma; metastatic; head and neck cancer; solid tumor; adoptive cell therapy; autologous; locally advanced refractory/recurrent melanoma; locally advanced refractory/recurrent head and neck cancer; IL-2
MeSH Terms: conditions — Melanoma; Head and Neck Neoplasms; Neoplasm Metastasis | interventions — Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Solid Tumor (Experimental): Solid Tumor
  Interventions: Biological: Autologous Tumor Infiltrating Lymphocytes; Biological: High-Dose Interleukin 2

INTERVENTIONS:
Biological: Autologous Tumor Infiltrating Lymphocytes — Autologous TILs
Biological: High-Dose Interleukin 2 — 720,000 IU/kg every 8 hours for up to 15 doses

SUMMARY:
To determine whether special tumor fighting cells that is taken from participants' tumors and grown in the laboratory and then given back to the participant will fight the participant's cancer when their immune system is suppressed from attacking these special tumor fighting cells.

DETAILED DESCRIPTION:
To determine whether special tumor fighting cells that is taken from participants' tumors and grown in the laboratory and then given back to the participant will fight the participant's cancer when their immune system is suppressed from attacking these special tumor fighting cells. This is called transfer of autologous (they came from you) tumor infiltrating lymphocytes (the cells that have been grown in the laboratory. Participants getting these cell infusions will also be treated with interleukin-2 (IL-2).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of head and neck squamous cell carcinoma OR metastatic cutaneous or mucosal melanoma measurable per RECIST.
* Progressive squamous cell cancer of the head and neck or metastatic melanoma since prior systemic treatment and who are:

  1. Not candidates for known curative intent therapy.
  2. Progressed following at least one prior systemic therapy.
  3. Have advanced melanoma unresectable stage III or stage IV
  4. Have advanced head and neck recurrent or metastatic disease
* Have no more than 3 brain metastases. Note: If lesions are symptomatic or ≥ 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
* Life expectancy of greater than 3 months.
* ECOG Performance Status of 0 or 1.
* Adequate organ and marrow function
* Seronegative for HIV antibody.
* Seronegative for Hepatitis B antigen, or Hepatitis C antibody or antigen.
* More than four weeks has elapsed since the patient received any prior systemic therapy at the time of enrollment.
* Patient has stable or progressing disease after at least one prior treatment.
* Six weeks or more have elapsed since the patient received any prior anti-CTLA4 antibody therapy

Exclusion Criteria:

* Currently using investigational agents.
* Had prior cell transfer therapy which included a non-myeloablative or myeloablative chemotherapy regimen.
* Patient is a female of child-bearing potential who is pregnant or breastfeeding
* Patient requires immune suppressive therapy including but not limited to greater than physiologic steroid replacement.
* Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Patient has any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
* Patient has opportunistic infections.
* Patient has a history of coronary revascularization or ischemic symptoms.
* Patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Daniels, MD, PhD, Principal Investigator — University of California, San Diego; Ezra Cohen, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Solid Tumor
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Solid Tumor
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Dose Limiting Toxicity (DLT)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Solid Tumor
Number analyzed (Participants) | 3
Participants
  Blood and Lymphatic System Disorders | 1
  Immune System Disorders, Renal and Urinary Disorders | 1
  Infections and Infestations, Endocrine Disorders, Metabolism and Nutrition Disorders, Investigations | 1

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Solid Tumor
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor (N=3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solid Tumor (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal re ux disease (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (5)
Bacteremia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT03991741/Prot_SAP_000.pdf